CLINICAL TRIAL: NCT03989986
Title: Peer-to-Peer (iP2P) Mentoring Program for Youth With Sickle Cell Disease: A Pilot Feasibility Randomized Controlled Trial
Brief Title: iPeer2Peer Program for Youth With Sickle Cell Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other); Royal University Hospital Foundation (Other); Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Senior Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1727
Record Dates: First submitted 2019-06-17; First posted 2019-06-18 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPeer2Peer Mentorship (Experimental): In addition to standard care, participants in the experimental group will receive the iPeer2Peer program, a peer mentorship program that will provide modelling and reinforcement of self-management by pre-screened and trained peer mentors (young adults with SCD aged 19-25 who have learned to function successfully with their condition). Mentors will encourage participants to develop and engage in self-management skills and provide social support.
  Interventions: Behavioral: iPeer2Peer Mentorship
- Waitlist Control Group (No Intervention): The control group participants will receive standard care and will be on a waitlist to receive the iPeer2Peer program until 15 weeks after completing their baseline questionnaires.

INTERVENTIONS:
Behavioral: iPeer2Peer Mentorship — Mentors and participants can have up to ten Skype calls over the course of 15 weeks.
  Arms: iPeer2Peer Mentorship

SUMMARY:
The iPeer2Peer Sickle Cell Disease (SCD) study matches youth (12-18 years of age) with SCD to a mentor (trained young adult) who has learned to manage their SCD well, transitioned to adult care, and can support youth participants emotionally and socially. Participants will be randomly assigned one of two groups, either (1) The intervention group: Study group participants are matched with a mentor for 15 weeks, and are expected to have up to ten calls with one another; (2) The control group: This study group will be on a 15 week waitlist to receive a mentor. This study will first assess the feasibility of conducting this research with youth with SCD. Also, this study will assess the preliminary effectiveness of peer mentorship by comparing various health outcomes of the two study groups post-intervention.

DETAILED DESCRIPTION:
Sickle Cell Disease (SCD) is a disease affecting red blood cells, where severe pain can develop due to blockage of red blood cells. This the most common genetic blood disease in North America, affecting mostly people of African descent. This type of pain can affect many aspects of one's life, and one's quality of life. Young people with SCD experience pain as they grow from childhood to adulthood, and experience daily chronic pain. There are many negative consequences of SCD, such as anxiety, depression, poor sleep, high stress, and limited social and physical activity. Peer support is a form of support that can provide someone with emotional, informational and social support. Peer support is a promising way of delivering emotional support, while helping someone learn how to cope and manage their disease. This is especially important for chronic diseases such as SCD, because young people will have to learn how to cope and manage their condition while growing up, and for the rest of their lives. A new way to provide face-to-face peer support is through the use of a virtual program using Skype via the Internet (to maintain face-to-face contact between mentors and mentees).

In this program, a young adult (a mentor) with a chronic disease is matched with a younger person living with the same disease (a mentee) online, through Skype. The mentors are nominated by their healthcare teams, and have successfully transitioned to adult care. They are trained to talk to young people about their disease and can give them some advice on how to manage, and grow up with the condition. This program has been tested with other groups with Juvenile Idiopathic Arthritis and Chronic Pain. A mentor and a mentee are matched for 15 weeks and are encouraged to have up to ten Skype calls together. The investigators do not know how well this program will work with young people with SCD. Therefore, the investigators would like to test out this program to see if it is feasible to conduct the iPeer2Peer SCD program in the future as a larger study with the SCD population.

Feasibility will be measured through the following: (1) recruitment and withdrawal rates; (2) rate of completion of weekly calls; (3) rate of completion of baseline measures; (4) estimates of intervention effects on health outcomes to inform the calculation of an appropriate sample size for the future definitive multi-centred randomized controlled trial (RCT) and (5) participants' perception regarding the acceptability of the SCD iP2P program and their level of engagement with the program (via a semi-structured interview). Descriptive statistics will be used to describe the sample characteristics at baseline. Rates of accrual, drop out, compliance, and missing data with 95% confidence intervals will be calculated.To inform sample size calculations and data analysis feasibility for a larger trial, data will be analyzed as in a larger study, and estimates of variance will be calculated. Secondary analysis will be conducted using an intent-to-treat approach. If assumptions for parametric statistics are met, linear regression models will be used to test intervention effects on pain impact, social support, self-efficacy, adherence and HRQL outcomes using an analysis of covariance approach with post-intervention measures compared between groups using baseline scores as covariates. The semi-structured individual (mentees) and focus group (mentors) interviews will determine (i) mentees' acceptability of and level of engagement in the iP2P program and (ii) mentors' likes and dislikes of program, improvement. This data, and subsequent analyses, will be used to refine the iP2P program prior to a full trial. A larger study will help to understand if peer support delivered by a mentor over Skype will help teenagers with SCD better manage their SCD, improve their health outcomes, and ultimately improve their quality of life living with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-18 years old
* Diagnosed with SCD by a haematologist
* Able to speak and read English
* Access to Internet connection with computer capable of using free Skype software
* Willing and able to complete online measures.

Exclusion Criteria:

* Significant cognitive impairments
* Major co-morbid illnesses (medical or psychiatric conditions) likely to influence HRQoL assessment
* Currently participating in other peer support or self-management interventions.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 2 years
  The number of participants recruited for the study during the recruitment study period.
Rates of completion of mentor-mentee calls | 15 weeks
  Compliance defined as 100% when a participant completes 10 calls within 15 weeks with their mentor
Withdrawal Rate | 2 years
  Number of participants that withdraw from the study over the study period
Acceptability of iPeer2Peer SCD intervention | 15 weeks
  Participants' perception regarding the acceptability of the SCD iP2P program and their level of engagement with the program (via a semi-structured interview).

SECONDARY OUTCOMES:
Sickle Cell Disease Pain Burden Interview- Youth | Baseline and 15 weeks after baseline completion.
  7-item questionnaire, measuring pain burden
Sickle Cell Disease Self-Efficacy Scale | Baseline and 15 weeks
  9-item questionnaire, measuring self-efficacy
PROMIS- Pediatric Peer Relationships 8a | Baseline and 15 weeks
  8-item questionnaire, measuring social support from peers
PROMIS depressive symptoms - 8a | Baseline and 15 weeks
  8-item questionnaire, measuring depression
PROMIS anxiety - 8a | Baseline and 15 weeks
  8-item questionnaire, measuring anxiety
PROMIS Pain Interference - 8a | Baseline and 15 weeks
  8-item questionnaire, measuring consequences of pain on relevant aspects of person's life.
PROMIS pain intensity - 1a | Baseline and 15 weeks
  1-item questionnaire, measuring intensity of pain over the past week
Transition-Q | Baseline and 15 weeks
  14-item questionnaire, measuring self-management

CONTACTS AND LOCATIONS:
Locations (4):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States
- Canada (3):
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Jim Pattison, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Lalji R, Koh L, Francis A, Khalid R, Guha C, Johnson DW, Wong G. Patient navigator programmes for children and adolescents with chronic diseases. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD014688. doi: 10.1002/14651858.CD014688.pub2. PMID 39382077